CLINICAL TRIAL: NCT06918288
Title: Post-extubation Support Using Nasal Humidified High-flow Oxygen Versus Non-invasive Positive Pressure Mechanical Ventilation in Preventing Reintubation Among Patients With Type II Respiratory Failure
Brief Title: Post-extubation Nasal Humidified High-flow Oxygen Versus Non-invasive Positive Pressure Ventilation
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Amr Tarek Atwa Heikal, Dr, Benha University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MD4-2-2025
Record Dates: First submitted 2025-03-15; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Respiratory Failure With Hypercapnia
Keywords: Difficult weaning-hypoxia-hypercapnea-postextubation-reintubation

STUDY DESIGN:
Intervention Model Description: To apply postextubation NIV or HFNC to prevent reintubation
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High flow nasal canula (HFNC) group. (Active Comparator)
  Interventions: Device: High flow nasal canula
- Non-invasive positive pressure mechanical ventilation (NIPPV) group. (Active Comparator)
  Interventions: Device: Non-invasive positive pressure mechanical ventilation

INTERVENTIONS:
Device: High flow nasal canula — All patients assigned to the HFNC group will receive HFNC immediately after extubation. Researchers will need to choose the suitable size nasal catheter. The initial airflow will be set to 50 L/min and adjusted according to patient tolerance with an absolute humidity setting to 44 mgH2O/L and the temperature setting to 37 °C.The patient's respiratory rate will be maintained below 30 beats/min or the baseline level before extubation with a SpO2 at 88-92%. HFNC failure is defined as escalation to NIV or invasive mechanical ventilation due to respiratory failure.
  Arms: High flow nasal canula (HFNC) group.
Device: Non-invasive positive pressure mechanical ventilation — All patients assigned to the control group will receive NIV immediately after extubation. Researchers will use a standard oronasal mask to connect the patient to the ventilator. The patients will be on Spontaneous/Timed (S/T) mode, with the initial end-expiratory pressure setting to 4 cmH2O. The pressure level will gradually increase to ensure that the patients can trigger the ventilator with each inhalation. The initial inspiratory pressure will be set at 8 cmH2O and adjusted according to the tidal volume with 6-8 ml/kg and tolerance of patients. The pres- sure level and the fraction of inspiration oxygen will be adjusted in order to maintain the respiratory rate ≤ 30/ min or the baseline level before extubation, a partial pressure of carbon dioxide (PaCO2) at 45-60 mmHg or the last PaCO2 level recorded before extubation, and a pulse oxygen saturation at 88-92%. NIV treatment failure is defined as a return to invasive mechanical ventilation.
  Arms: Non-invasive positive pressure mechanical ventilation (NIPPV) group.

SUMMARY:
Acute hypercapnic respiratory failure (AHRF), which is commonly defined as arterial partial pressure of carbon dioxide (PaCO2) ≥ 45 mmHg and frequently accompanied by reduced levels of arterial partial pressure of oxygen (PaO2), can occur in a variety of etiologies, mainly in chronic respiratory diseases, such as exacerbation of chronic obstructive pulmonary disease, cystic fibrosis, thoracic deformities, as well as other conditions, such as neuromuscular disease The purpose of this research is to To compare efficacy of administration of high flow nasal canula versus non-invasive mechanical ventilation on preventing reintubation during 72 hours postextubation of patients with type 2 respiratory failure with difficult weaning.

ELIGIBILITY:
Inclusion Criteria:

* The study will be recruited on type II respiratory failure patients with difficult weaning from invasive mechanical. Patients who will fulfil the eligibility criteria will be randomly divided into HFNC or NIV groups to receive sequential treatment after extubation.

Hypercapnic respiratory failure is defined as an elevation in PaCO2 greater than 45 mmHg and a pH lower than 7.35 resulting from respiratory pump failure and/or production.

Type 2 respiratory failure common causes :

1. Neuromuscular Disorders such as: Amyotrophic lateral sclerosis (ALS), Myasthenia gravis, Muscular dystrophy.
2. Spinal cord injuries or damage to the spinal cord that can impair respiratory function.
3. Pulmonary Disorders Like Chronic obstructive pulmonary disease (COPD) ,Cystic fibrosis, Pneumonia Severe infection can cause respiratory failure , Pulmonary embolism.
4. Obesity and Sleep-Related Disorders like Obesity hypoventilation syndrome (OHS), obstructive sleep apnea(OSA).
5. Chest Wall and Pleural Disorders as Kyphoscoliosis, Pleural effusion, Pneumothorax.
6. Other Causes: Sedative overdose, Neurological disorders, high altitude

Exclusion Criteria:

* 1. Lack of informed consent. 2. A contraindication to NIV (oral and facial trauma, excessive phlegm with poor expectoration ability, hemodynamic instability, recent esophageal surgery).

  3. Patients with poor short-term prognosis (very high risk of death within seven days or receiving palliative care).

  4. Other organs' failure e.g severe heart, brain, liver, or kidney failure. 5. Tracheostomised patients. 6. Loss of follow up and uncertain 28 day survival.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
The primary outcomes of this study will be the rate of re- intubation | 72 hours and 7 days after extubation.
  frequency of re-intubation

SECONDARY OUTCOMES:
ventilator-free days | 28 days post-randomization
  ventilator-free days at 28 days post-randomization
duration of respiratory support after extubation. | 72 hours after extubation
  duration of respiratory support after extubation
treatment failure and reintubation rate | during 48 hours after extubation.
  treatment failure rate (including reintubation rate and replacement of respiratory support: for patients in the HFNC group, treatment failure means to upgrade to NIV or invasive mechanical ventilation; for patients in the NIV group, treatment failure means to change to invasive mechanical ventilation).
respiratory support related adverse events | 72 hours post extubation
  respiratory support related adverse events
Delirium | 72 hours postextubation
  the incidence of delirium using RAAS (Richmond Agitation-sedation score)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Mostafa Abdelhamid, Professor of Anesthesia, Study Director — faculty of medicine, Benha university; Fatma Ahmed Abdelfattah, MD Anesthesia and intensive ca, Principal Investigator — faculty of medicine, Benha university; Mohamed Shaker Sadek, MD chest diseases, Study Chair — faculty of medicine, Benha university
Locations (1):
- Banha Faculity of Medicine, Banhā, Elqalyoubea, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Thille AW, Harrois A, Schortgen F, Brun-Buisson C, Brochard L. Outcomes of extubation failure in medical intensive care unit patients. Crit Care Med. 2011 Dec;39(12):2612-8. doi: 10.1097/CCM.0b013e3182282a5a. PMID 21765357
- [Background] Comellini V, Pacilli AMG, Nava S. Benefits of non-invasive ventilation in acute hypercapnic respiratory failure. Respirology. 2019 Apr;24(4):308-317. doi: 10.1111/resp.13469. Epub 2019 Jan 12. PMID 30636373
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30636373/
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/21765357/
- Available data/document: Clinical Study Report: Arnaud W Thille et al — http://pubmed.ncbi.nlm.nih.gov/21765357/ — Extubation failure is associated with a poor prognosis, but the respective roles for reintubation per se and underlying disease severity remain unclear. Our objectives were to evaluate the impact of failed extubation, whether planned or unplanned, on patient outcomes and to identify a patient subset at risk for extubation failure.